CLINICAL TRIAL: NCT03145779
Title: Evaluation of Phenotypic Variability in Fabry Disease
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Farrah Rajabi, Instructor, Division of Genetics and Genomics, Boston Children's Hospital
Other Study IDs: IRB-P00022060
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebrovascular events, such as stroke, are a devastating complication of Fabry disease that results in part from storage of complex lipids in both large and small vessels. Understanding how the genotype influences the phenotype or clinical presentation can help us understand which patients are at risk for the complications of Fabry disease. This study aims to follow the natural history of this disease will help us understand and predict long-term outcomes for patients.

DETAILED DESCRIPTION:
This longitudinal study will be conducted at Boston Children's Hospital (BCH). Subjects recruited for the study will have routine clinical care assessment with a complete physical and neurological exam and biochemical monitoring with venipuncture. In addition as part of the study, subjects will be given questionnaires to assess details of medical and psychosocial history, will complete self-reported measures of neuropsychological evaluation, pain scores, quality of life, executive functioning and cognitive functioning. All patients assessments will be repeated every 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who carry a classic alpha-galactosidase gene (GLA) mutation
* All ages
* Medical records available including previous genetic testing.
* Capable of providing informed consent with assent for patients less than 18 years
* Not currently involved in any other clinical trials.

Exclusion Criteria:

* No medical records available
* No record of genotype
* Not capable of providing informed consent
* Currently involved in any clinical trial

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of Fabry disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Globotriaosylceramide level, plasma | Data will be obtained and studied every 2 years for up to 10 years.
  Biomarker for deficiency of alpha-galactosidase A (GLA) activity measured to determine if there are changes over time.
Globotriaosylceramide level, urine | Data will be obtained and studied every 2 years for up to 10 years.
  Biomarker for deficiency of alpha-galactosidase A (GLA) activity measured to determine if there are changes over time.
Intelligence scale assessment | Data will be obtained and studied every 2 years for up to 10 years.
  Wechsler Adult Intelligence Scale - Revised (WAIS-R) to assess for any changes in intelligence scale over time.
Quality of life questionnaire | Data will be obtained and studied every 2 years for up to 10 years.
  Single score based on questionnaire about quality of life to assess for any changes in scores over time.
Executive functioning test | Data will be obtained and studied every 2 years for up to 10 years.
  Single score based on testing of digit span backwards test, letter fluency, and category fluency to assess any changes in executive function over time.
Pain questionnaire | Data will be obtained and studied every 2 years for up to 10 years.
  Single score based on questionnaire about pain to evaluate progression of pain scores over time.
Physical exam | Data will be obtained and studied every 2 years for up to 10 years.
  Physical exam to evaluate for the development of angiokeratoma lesions and neurological symptoms development over time.

SECONDARY OUTCOMES:
Transcriptome analysis | Data will be obtained and studied every 2 years for up to 10 years.
  High-throughput RNA sequencing will be done on plasma and peripheral blood lymphocytes to evaluate for changes over time.
Metabolomic analysis | Data will be obtained and studied every 2 years for up to 10 years.
  Comprehensive metabolite mapping of biochemical pathways to determine any metabolomic pathway changes in Fabry disease patients over time.
Microbiome analysis | Data will be obtained and studied every 2 years for up to 10 years.
  Optional stool sample will be obtained for microbiome analysis to detect the microbiome progression over time in Fabry disease patients.
Targeted exome sequencing for evaluation of potential modifiers of Fabry disease phenotype. | Data will be obtained one time at initial study visit
  Investigators will analyze sequencing results to determine the ability of whole exome sequencing to detect pathogenic modifiers of the Fabry disease phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No